CLINICAL TRIAL: NCT04761458
Title: Correlation of Preoperative Global Olfactory Function With Frailty, Preoperative Cognitive Status, Postoperative Neurocognitive Disorders and Mortality Following Elective Surgery
Brief Title: Correlation of Preoperative Global Olfactory Function With Frailty, Perioperative Neurocognitive Disorders and Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: B403202043093
Record Dates: First submitted 2021-02-03; First posted 2021-02-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Perioperative/Postoperative Complications; Olfactory Disorder; Neurocognitive Disorders; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Frailty; Postoperative Complications; Neurocognitive Disorders; Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled for elective surgery aged 65 and + (Experimental)
  Interventions: Diagnostic Test: Olfactory function testing; Diagnostic Test: Edmonton Frail Scale; Diagnostic Test: Clinical Frailty Scale; Diagnostic Test: Neuropsychological test battery

INTERVENTIONS:
Diagnostic Test: Olfactory function testing — Olfactory function will be evaluated through the Burghart Sniffin' Sticks test which is a validated psychophysical testing method. Sniffin' Sticks test is based on pen-like odor dispensing devices that will be presented to the patients. The extended version of this test will be used and consist of three tests of olfactory function, namely tests for odor threshold, odor discrimination and odor identification.
Diagnostic Test: Edmonton Frail Scale — The Edmonton Frail Scale (EFS) involves nine domains of frailty : functional performance, cognitive function, general health, functional independence, social support, used medications, nutrition, mood and continence. It has been validated with respect to comprehensive geriatric assessment and to other screening tools related to frail state. EFS test is considered most appropriate for use in routine preoperative screening and only requires 5 minutes.
Diagnostic Test: Clinical Frailty Scale — The Clinical Frailty Scale (CFS) uses clinicians' judgement to evaluate frailty. It comprises assessment of specific domains including comorbidity, function, and cognition. Score ranges from 1 (very fit) to 9 (terminally ill).
Diagnostic Test: Neuropsychological test battery — Patients will undergo a neuropsychological test battery preoperatively and postoperatively. This test consists of a battery of psychometric assessments with the ability to objectively assess specific cognitive domains such as attention, executive function, learning and memory, language, perceptual-motor, or social cognition.

SUMMARY:
The aims of this research project are to evaluate whether global olfactory impairment is a reliable indicator of preoperative frailty and cognitive impairment, and whether it may predict postoperative neurocognitive disorders, morbidity and mortality in a population of older patients scheduled for elective intermediate- to high-risk elective surgery.

1. We will measure preoperative global olfactory function (threshold, discrimination, identification) and evaluate whether olfactory impairment predicts preoperative frailty (using the Edmonton Frail Scale, the Clinical Frailty Scale and handgrip strength) and postoperative complications and mortality.
2. We will address the question whether preoperative olfactory impairment may be associated with a preoperative cognitive impairment (through a neuropsychological test battery) and whether it may predict a decrease in postoperative neurocognitive function.

DETAILED DESCRIPTION:
Olfactory impairment increases with age, affecting more than 50% of the population aged between 65 and 80 years old. Recently, many studies have demonstrated a strong association between olfactory impairment and overall mortality risk. At the moment, the underlying physiopathology linking olfactory impairment to mortality remains unknown and only putative mechanisms are suggested.

Among them, accelerated physiological brain aging seems to be involved, making olfactory decline a possible marker of frailty. To date, only a few studies (mostly using subjective olfactory assessment) investigated the potential relationship between olfactory impairment and frailty. Moreover, neurodegenerative diseases, through cognitive dysfunction, seem likely to represent a second mechanism potentially underlying the link between olfactory impairment and mortality.

Surgery, and more broadly the perioperative period, remains a major source of morbidity and mortality. Meanwhile, the average age of the surgical population continues to rise, making preoperative risk assessment an essential step in order to detect the most vulnerable patients. Yet, it is well-known that frailty is predictive of complications and mortality and that preoperative cognitive impairment is associated with postoperative neurocognitive disorders.

The first objective of this research project is thus to evaluate global olfactory function of preoperative older surgical patients in light of an assessment of their frailty and cognitive status. Frailty will be tested with the Edmonton Frail Scale, the Clinical Frailty Scale and handgrip strength. Cognitive function will be tested through a neuropsychological test battery preoperatively and postoperatively. The second and third objectives are to correlate preoperative olfactory function with, on the one hand, postoperative neurocognitive disorders, and on the other hand, postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery (covering orthopedic, spine and cardiovascular surgery)

Exclusion Criteria:

* History of neurological or psychiatric disorder
* History of severe head trauma
* History of olfactory trouble or chronic rhinosinusitis or sinus surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 215 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of frailty assessed by the Edmonton Frail Scale | Preoperative period (within 3 months before surgery)
  Analysis of the prevalence of frailty assessed by the Edmonton Frail Scale according to preoperative olfactory function (Burghart Sniffin' Sticks extended test).
Prevalence of frailty assessed by the Clinical Frailty Scale | Preoperative period (within 3 months before surgery)
  Analysis of the prevalence of frailty assessed by the Clinical Frailty Scale according to preoperative olfactory function (Burghart Sniffin' Sticks extended test).
Incidence of postoperative complications | Up to 1 year postoperatively
  Analysis of the incidence of postoperative complications according to preoperative olfactory function (Burghart Sniffin' Sticks extended test).
Incidence of mortality | Up to 1 year postoperatively
  Analysis of the incidence of mortality according to preoperative olfactory function (Burghart Sniffin' Sticks extended test).

SECONDARY OUTCOMES:
Prevalence of preoperative neurocognitive disorder | Preoperative period (within 3 months before surgery)
  Analysis of the prevalence of neurocognitive disorder (assessed through a neuropsychological test battery) according to preoperative olfactory function.
Incidence of postoperative neurocognitive disorder | From 6 weeks to 12 weeks postoperatively
  Analysis of the incidence of postoperative neurocognitive disorder (assessed through a neuropsychological test battery) according to preoperative olfactory function.

OTHER OUTCOMES:
Postoperative global olfactory function (Burghart Sniffin' Sticks extended test) | From 6 weeks to 12 weeks postoperatively
  Comparison of preoperative and postoperative global olfactory function (both assessed through Burghart Sniffin' Sticks extended test)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Van Regemorter, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Pinto JM, Wroblewski KE, Kern DW, Schumm LP, McClintock MK. Olfactory dysfunction predicts 5-year mortality in older adults. PLoS One. 2014 Oct 1;9(10):e107541. doi: 10.1371/journal.pone.0107541. eCollection 2014. PMID 25271633
- [Background] Schubert CR, Fischer ME, Pinto AA, Klein BEK, Klein R, Tweed TS, Cruickshanks KJ. Sensory Impairments and Risk of Mortality in Older Adults. J Gerontol A Biol Sci Med Sci. 2017 May 1;72(5):710-715. doi: 10.1093/gerona/glw036. PMID 26946102
- [Background] Van Regemorter V, Hummel T, Rosenzweig F, Mouraux A, Rombaux P, Huart C. Mechanisms Linking Olfactory Impairment and Risk of Mortality. Front Neurosci. 2020 Feb 21;14:140. doi: 10.3389/fnins.2020.00140. eCollection 2020. PMID 32153360
- [Background] Somekawa S, Mine T, Ono K, Hayashi N, Obuchi S, Yoshida H, Kawai H, Fujiwara Y, Hirano H, Kojima M, Ihara K, Kim H. Relationship between Sensory Perception and Frailty in a Community-Dwelling Elderly Population. J Nutr Health Aging. 2017;21(6):710-714. doi: 10.1007/s12603-016-0836-5. PMID 28537337
- [Background] Laudisio A, Navarini L, Margiotta DPE, Fontana DO, Chiarella I, Spitaleri D, Bandinelli S, Gemma A, Ferrucci L, Incalzi RA. The Association of Olfactory Dysfunction, Frailty, and Mortality Is Mediated by Inflammation: Results from the InCHIANTI Study. J Immunol Res. 2019 Feb 20;2019:3128231. doi: 10.1155/2019/3128231. eCollection 2019. PMID 30915369
- [Background] Harita M, Miwa T, Shiga H, Yamada K, Sugiyama E, Okabe Y, Miyake Y, Okuno T, Iritani O, Morimoto S. Association of olfactory impairment with indexes of sarcopenia and frailty in community-dwelling older adults. Geriatr Gerontol Int. 2019 May;19(5):384-391. doi: 10.1111/ggi.13621. Epub 2019 Apr 9. PMID 30968523